CLINICAL TRIAL: NCT01521832
Title: A Phase I, Randomised, Double-Blind, Placebo-Controlled, Two-Part Study Consisting of Single and Multiple Oral Dose Escalation to Determine, Safety, Tolerability and Pharmacokinetics of SEN0014196
Brief Title: Escalating Dose Study in Healthy Volunteers With SEN0014196
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Siena Biotech S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: S015-001
Record Dates: First submitted 2012-01-13; First posted 2012-01-31 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-01

CONDITIONS: Huntington's Disease
MeSH Terms: conditions — Huntington Disease | interventions — 6-chloro-2,3,4,9-tetrahydro-1H-carbazole-1-carboxamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (11):
- Dose Group A (Experimental)
  Interventions: Drug: SEN0014196
- Dose Group B (Experimental)
  Interventions: Drug: SEN0014196
- Dose Group C (Experimental)
  Interventions: Drug: SEN0014196
- Dose Group D (Experimental)
  Interventions: Drug: SEN0014196
- Dose Group E (Experimental)
  Interventions: Drug: SEN0014196
- Dose Group F (Experimental)
  Interventions: Drug: SEN0014196
- Dose Group H (Experimental)
  Interventions: Drug: SEN0014196
- Dose Group I (Experimental)
  Interventions: Drug: SEN0014196
- Dose Group J (Experimental)
  Interventions: Drug: SEN0014196
- Dose Group K (Experimental)
  Interventions: Drug: SEN0014196
- Dose Group L (Experimental)
  Interventions: Drug: SEN0014196

INTERVENTIONS:
Drug: SEN0014196 — 5 mg single oral dose
  Arms: Dose Group A
Drug: SEN0014196 — 25 mg single oral dose
  Arms: Dose Group B
Drug: SEN0014196 — 75 mg single oral dose
  Arms: Dose Group C
Drug: SEN0014196 — 150 mg single oral dose
  Arms: Dose Group D
Drug: SEN0014196 — 300 mg single oral dose
  Arms: Dose Group E
Drug: SEN0014196 — 600 mg single oral dose
  Arms: Dose Group F
Drug: SEN0014196 — 300 mg single oral dose (females)
  Arms: Dose Group H
Drug: SEN0014196 — 100 mg multiple oral dose
  Arms: Dose Group I
Drug: SEN0014196 — 300 mg multiple oral dose
  Arms: Dose Group J
Drug: SEN0014196 — 100 mg BID multiple oral dose
  Arms: Dose Group K
Drug: SEN0014196 — 100 mg BID multiple oral dose (females)
  Arms: Dose Group L

SUMMARY:
This is a trial in healthy volunteers to study the safety, tolerability and pharmacokinetics of single and multiple escalating doses of SEN0014196.

ELIGIBILITY:
Inclusion Criteria:

* Subjects in Groups A to G and Groups I to K will be males of any ethnic origin between 18 and 55 years of age and with a body mass index (BMI) between 18 and 31 kg/m2 inclusive. Subjects in Groups H and L will be females of any ethnic origin between 18 and 65 years of age and with a body mass index (BMI) between 18 and 31 kg/m2 inclusive. All subjects will have a body weight greater than 50 kg. For Group H, women will be of non-childbearing potential, defined as follows: Female subjects 50 years of age or less must be surgically sterile or post-menopausal (defined as at least two years post cessation of menses and/or follicular stimulating hormone >18 mIU/mL and serum oestradiol <110 pmol/L), non-lactating and have a negative serum pregnancy test Female subjects of more than 51 years of age must be surgically sterile or post-menopausal (defined by a value of follicular stimulating hormone >18 mIU/mL and no spontaneous menstruation for at least one year before the first dose), non-lactating and have a negative serum pregnancy test.
* Subjects must be in good health, as determined by a medical history, physical examination, 12-lead electrocardiogram (ECG) and clinical laboratory evaluations Note: congenital non-haemolytic hyperbilirubinaemia is not acceptable and serum potassium must be within the normal reference ranges (confirmed by repeat analysis).
* Subjects will have given their written informed consent to participate in the study and to abide by the study restrictions.

Exclusion Criteria:

* Male subjects or Female subjects in Group H who are not, or whose partners are not willing to use appropriate contraception (such as condom) with spermicidal foam/gel/film/cream/suppository) from the time of the first dose until 3 months after the final dosing occasion. Female subjects in Group L who are not, willing to use appropriate contraception (such as condom) with spermicidal foam/gel/film/cream/suppository) from the time of screening until 3 months after the final dosing occasion, who have not had a menstrual period in the 28 days before the first dose.
* Subjects who have received any prescribed systemic or topical medication within 14 days of the first dose administration (for female subjects, stable hormone replacement therapy is acceptable) unless in the opinion of the Investigator the medication will not interfere with the study procedures or compromise safety.
* Subjects who have used any non-prescribed systemic or topical medication (including herbal remedies) within 7 days of the first dose administration (with the exception of vitamin/mineral supplements) unless in the opinion of the Investigator the medication will not interfere with the study procedures or compromise safety.
* Subjects who have received any medications, including St John's Wort, known to chronically alter drug absorption or elimination processes within 30 days of the first dose administration unless in the opinion of the Investigator the medication will not interfere with the study procedures or compromise safety
* Subjects who are still participating in a clinical study (e.g. attending follow-up visits) or who have participated in a clinical study involving administration of an investigational drug (new chemical entity) in the past 3 months, where possible this will be confirmed using The Over Volunteering Protection Service (TOPS).
* Subjects who have donated any blood, plasma or platelets in the 2 months prior to screening or who have made donations on more than two occasions within the 12 months preceding the first dose administration.
* Subjects with a significant history of drug allergy as determined by the Investigator.
* Subjects who have any clinically significant allergic disease (excluding non-active hayfever) as determined by the Investigator.
* Subjects who have a supine blood pressure and supine pulse rate higher than 140/90 mmHg and 100 beats per minute (bpm), respectively, or lower than 90/50 mmHg and 40 bpm, respectively, confirmed by a repeat assessment.
* Subjects who consume more than 28 units (males) or more than 21 units (females) of alcohol per week or who have a significant history of alcoholism or drug/chemical abuse as determined by the Investigator (one unit of alcohol equals ½ pint [285 mL] of beer or lager, one glass [125 mL] of wine, or 1/6 gill [25 mL] of spirits).
* Subjects with a positive urine drug screen or alcohol breath test result at screening or first admission. Or a history of substance abuse in the last 12 months prior to the start of the study.
* Subjects who smoke more than 5 cigarettes or the equivalent in tobacco per day.
* Subjects with, or with a history of, any clinically significant neurological, gastrointestinal, renal, hepatic, cardiovascular, psychiatric, respiratory, metabolic, endocrine, haematological or other major disorders as determined by the Investigator.
* Subjects with, or with a family history of Huntington's Disease
* Subjects who have previously received histone deacetylase inhibitors e.g. vorinostat (Zolinza®) or have participated in a clinical trial using a histone deacetylase inhibitor.
* Subjects who have had a clinically significant illness within 4 weeks of the start of dose administration as determined by the Investigator
* Subjects who are known to have serum hepatitis, or who are carriers of the hepatitis B surface antigen (HBsAg) or hepatitis C antibody, or who have a positive result to the test for HIV antibodies.
* Subjects who have an abnormality in the 12-lead ECG that, in the opinion of the investigator, increases the risk of participating in the study, such as QTcF interval >450 msec (male) or greater than 470msec (female), or with sinus rhythm with PR interval <110 msec or >240 msec, confirmed by a repeat ECG.
* Subjects who, in the opinion of the Investigator, should not participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2009-10; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of ascending single and multiple oral doses of SEN0014196 in healthy male and female subjects. | Up to 7 days after single dose and up to 10 days following multiple dose
  Vital signs, cardiovascular and neurological function, laboratory safety parameters. Type and frequancy of adverse events.

SECONDARY OUTCOMES:
Single and multiple dose pharmacokinetics of SEN0014196 | Up to 96 hours following single dose and up to 48 hours following multiple dose.
  Basic pharmacokinetic parameters (Cmax, AUC, accumulation ratio, gender differences).

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Chiesa, MD, Principal Investigator — Covance
Locations (1):
- Covance Clinical Research Unit, Leeds, United Kingdom

REFERENCES:
- [Derived] Westerberg G, Chiesa JA, Andersen CA, Diamanti D, Magnoni L, Pollio G, Darpo B, Zhou M. Safety, pharmacokinetics, pharmacogenomics and QT concentration-effect modelling of the SirT1 inhibitor selisistat in healthy volunteers. Br J Clin Pharmacol. 2015 Mar;79(3):477-91. doi: 10.1111/bcp.12513. PMID 25223836